CLINICAL TRIAL: NCT01683240
Title: Prospective Multicenter Evaluation of a New Short-access-cholangioscope for Biliary Duct Strictures and Gall Stones
Acronym: SAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: KARL STORZ GmbH & Co. KG, Tuttlingen, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Short Access Cholangioscope; PV 3526 (Registry Identifier: Hamburg Ethical Committee)
Record Dates: First submitted 2012-07-06; First posted 2012-09-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Choledocholithiasis; Common Bile Duct Neoplasms; Cholestasis
Keywords: cholangiography; cholangioscopy; mother-baby; cholangioscope; Frimberger cholangioscope; short access cholangioscopy; ERCP; gallstone therapy
MeSH Terms: conditions — Choledocholithiasis; Common Bile Duct Neoplasms; Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Frimberger cholangioscope (Experimental): Patients with need for cholangioscopy due to gallstones or histological evaluation of strictures
  Interventions: Device: cholangioscopy (Frimberger)

INTERVENTIONS:
Device: cholangioscopy (Frimberger) — cholangioscopy with Frimberger duodenoscope system by the company of Karl Storz GmbH

SUMMARY:
Karl Storz GmbH (Gesellschaft mit beschränkter Haftung) company developed a cholangioscopic device, which is designed to give a better flexibility to the cholangioscopy tip in order to enable optimal diagnostic and therapeutic precondition. Other than the conventional mother-baby technique, the insertion of the cholangioscope (baby part) is done by a port at the side of a specially developed duodenoscope (mother part) which is prepositioned distally to the control unit, near to the patient's mouth. Better manoeuverability of the device tip will lead to both a better accuracy in taking biopsies as well as a better flexibility in lithotripsy manoeuvres. This study is designed to test the efficiency of the device in relation to this assumption.

DETAILED DESCRIPTION:
Cholangioscopy is a subsidiary treatment in endoscopic retrograde cholangiopancreaticography (ERCP), used for special issues. In the context of ERCP, a long,thin shaped device is introduced through the working channel of a duodenoscope and then through the papilla into the biliary duct.

Inspection of the biliary duct can be used for tumor biopsies as well as for gall stone lithotripsy by laser or electrohydraulic technique.

Manoeuverability of cholangioscopes is limited by the length of the scope, even more, since most of the device body is stuck in the working channel.

The newly designed cholangioscope by the company of Karl Storz GmbH is introduced through a shortened working channel. Introduction of the cholangioscope is done by an innovative side port for the cholangioscope at 70 cm from the insertion tube's distal end. This leads to a better flexibility of the device tip. Better manoeuverability of the device tip will lead to both a better accuracy in taking biopsies as well as a better flexibility in lithotripsy manoeuvres.

This study is designed to test the efficiency of the device in relation to this assumption.

ELIGIBILITY:
Inclusion Criteria:

* Choledocholithiasis, not treatable through conventional ERCP with sphincterotomy.
* Stricture of the biliary duct in need of histopathological investigation

Exclusion Criteria:

* Aggravated or impossible access to papilla
* Inappropriate biliary anatomy, e.g. multiple strictures or diameter of duct < cholangioscope impairing intubation
* Primary sclerosing cholangitis
* Coagulopathy (quick < 50%, thrombocytes < 50/nl)and anticoagulant medication
* Bad patient's condition (ASA IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of cholangioscopy in gallstone therapy and stricture diagnosis | Patients will be monitored during stay in hospital, average stay is 1 day
  1. complete lithotripsy in a single session
  2. rate of right positive malignoma diagnostics (sensitivity)

SECONDARY OUTCOMES:
Complication rate | while examination and 24 hrs past examination
  Number of complications during examination and during monitoring over 24 hours post procedure
Gallstone therapy | procedure, average procedure time 1 hour
  Time of procedure and success of stone extraction in %
Stricture diagnostic | procedure, average procedure time is 1 hour
  Number of biopsies taken. Evaluation of quality of biopsies by pathologists (pathological department of University Hospital Hamburg Eppendorf).
  Minimum number of bioptic manoeuvres: 3 Comparison with brush cytology (3 brush manoeuvres with 12 smear preparations) by reference cytologist (Dr. Topalidis, Hannover)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (5):
- Germany (5):
  - Charité Universitätsmedizin, Virchow Klinikum, Berlin
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Hamburg Barmbek, Hamburg
  - Israelitisches Krankenhaus, Hamburg
  - Asklepios Klinik Hamburg Altona, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pomerantz BJ. Biliary tract interventions. Tech Vasc Interv Radiol. 2009 Jun;12(2):162-70. doi: 10.1053/j.tvir.2009.08.009. PMID 19853234
- [Background] Tsuyuguchi T, Fukuda Y, Saisho H. Peroral cholangioscopy for the diagnosis and treatment of biliary diseases. J Hepatobiliary Pancreat Surg. 2006;13(2):94-9. doi: 10.1007/s00534-005-1064-2. PMID 16547668
- [Background] Ross AS, Kozarek RA. Cholangioscopy: where are we now? Curr Opin Gastroenterol. 2009 May;25(3):245-51. doi: 10.1097/MOG.0b013e328329236c. PMID 19381085
- [Background] Darcy M, Picus D. Cholangioscopy. Tech Vasc Interv Radiol. 2008 Jun;11(2):133-42. doi: 10.1053/j.tvir.2008.07.007. PMID 18922458
- [Background] Small AJ, Baron TH. Novel endoscopic approaches for assessing biliary tract diseases. Curr Opin Gastroenterol. 2008 May;24(3):357-62. doi: 10.1097/MOG.0b013e3282fad830. PMID 18408465
- [Background] Fukuda Y, Tsuyuguchi T, Sakai Y, Tsuchiya S, Saisyo H. Diagnostic utility of peroral cholangioscopy for various bile-duct lesions. Gastrointest Endosc. 2005 Sep;62(3):374-82. doi: 10.1016/j.gie.2005.04.032. PMID 16111955
- [Background] Kim HJ, Kim MH, Lee SK, Yoo KS, Seo DW, Min YI. Tumor vessel: a valuable cholangioscopic clue of malignant biliary stricture. Gastrointest Endosc. 2000 Nov;52(5):635-8. doi: 10.1067/mge.2000.108969. PMID 11060188
- [Background] Nimura Y, Kamiya J, Hayakawa N, Shionoya S. Cholangioscopic differentiation of biliary strictures and polyps. Endoscopy. 1989 Dec;21 Suppl 1:351-6. doi: 10.1055/s-2007-1012989. PMID 2606085
- [Background] Seo DW, Lee SK, Yoo KS, Kang GH, Kim MH, Suh DJ, Min YI. Cholangioscopic findings in bile duct tumors. Gastrointest Endosc. 2000 Nov;52(5):630-4. doi: 10.1067/mge.2000.108667. PMID 11060187
- [Background] Tamada K, Ueno N, Tomiyama T, Oohashi A, Wada S, Nishizono T, Tano S, Aizawa T, Ido K, Kimura K. Characterization of biliary strictures using intraductal ultrasonography: comparison with percutaneous cholangioscopic biopsy. Gastrointest Endosc. 1998 May;47(5):341-9. doi: 10.1016/s0016-5107(98)70216-0. PMID 9609424
- [Background] Itoi T, Sofuni A, Itokawa F, Tsuchiya T, Kurihara T, Ishii K, Tsuji S, Moriyasu F, Gotoda T. Peroral cholangioscopic diagnosis of biliary-tract diseases by using narrow-band imaging (with videos). Gastrointest Endosc. 2007 Oct;66(4):730-6. doi: 10.1016/j.gie.2007.02.056. PMID 17905015
- [Background] Hoffman A, Kiesslich R, Bittinger F, Galle PR, Neurath MF. Methylene blue-aided cholangioscopy in patients with biliary strictures: feasibility and outcome analysis. Endoscopy. 2008 Jul;40(7):563-71. doi: 10.1055/s-2007-995688. Epub 2008 Apr 11. PMID 18404601